CLINICAL TRIAL: NCT02425631
Title: CT Follow-Up of the SImmetry Sacroiliac Joint Fusion System
Status: Completed | Type: Observational
Sponsor: Zyga Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL1097
Record Dates: First submitted 2015-04-16; First posted 2015-04-24 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Sacroiliitis
Keywords: SI joint fusion; SI joint pain; SI joint; SI joint treatment; SI joint disease; Sacroiliac joint; Simmetry
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SImmetry Sacroiliac Joint Fusion System — Minimally invasive surgery for implantation of the SImmetry System

SUMMARY:
This study will evaluate long-term follow-up of subjects implanted with the SImmetry Sacroiliac (SI) Joint Fusion System (SImmetry).

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a SImmetry device implanted.
* Patient is willing to comply with study procedures and provide informed consent.

Exclusion Criteria:

* Patient is physically unable to return to the clinic for CT imaging.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with the SImmetry System will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
SI Joint Fusion (CT evidence of SI joint fusion) | 12 months
  CT evidence of SI joint fusion evaluated by a core laboratory

SECONDARY OUTCOMES:
SI Joint Pain (CT evidence of SI joint fusion) | 24 months
  evaluated by a core laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Ingham, Study Director — Zyga